CLINICAL TRIAL: NCT06735209
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 1 Trial to Evaluate the Safety, Tolerability, Immunogenicity, and Efficacy of Sanaria(R) PfSPZ-LARC2 Vaccine, a Late-Arresting, Replication-Competent, Genetically Attenuated Plasmodium Falciparum Vaccine by Controlled Human Malaria Infection in Malaria-Naïve Healthy Adults
Brief Title: First-in-Human PfSPZ-LARC2 Vaccination/CHMI
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 23-0010; 5UM1AI148684-04 (NIH)
Record Dates: First submitted 2024-11-22; First posted 2024-12-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-05-20

CONDITIONS: Malaria
Keywords: Artemether/lumefantrine (Coartem(R)); Atovaquone/proguanil (Malarone(R)); CHMI; controlled; First-in-human; Malaria; Plasmodium falciparum; Saline; Sanaria(R) PfSPZ Challenge (7G8); Sanaria(R) PfSPZ-LARC2; Sentinel; Vaccine
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Clinic Study Staff (except for Pharmaceutical Operations), Study Statistician and Lab staff will be unaware of the treatment group assignment. Products for administration will be indistinguishable to the participants, the persons administering vaccine, and persons conducting laboratory assays, and this blinding will be maintained by study staff for clinical evaluations thereafter until after the CHMI phase is completed.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Experimental): Healthy malaria-naïve participants aged between 18 and 45 years will receive 2x10^5 PfSPZ of Plasmodium falciparum sporozoite vaccine (PfSPZ-LARC2) vaccine on Days 1, 29, and 57 followed by 3.2x10^3 PfSPZ Challenge (7G8) Controlled Human Malaria Infection (CHMI) on Day 169 administered by direct venous inoculation (DVI). Placebo participants that drop out prior to CHMI will be replaced with infectivity controls. Infectivity controls will receive PfSPZ Challenge (7G8) CHMI N=3
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ (7G8) Challenge
- Group 2 (Placebo Comparator): Healthy malaria-naïve participants aged between 18 and 45 years will receive saline placebo on Days 1, 29, and 57 followed by 3.2x10^3 PfSPZ Challenge (7G8) Controlled Human Malaria Infection (CHMI) on Day 169 administered by direct venous inoculation (DVI). Placebo participants that drop out prior to CHMI will be replaced with infectivity controls. Infectivity controls will receive PfSPZ Challenge (7G8) CHMI N=1
  Interventions: Biological: PfSPZ (7G8) Challenge; Other: Sodium Chloride, 0.9%
- Group 3 (Experimental): Healthy malaria-naïve participants aged between 18 and 45 years will receive 2x10^5 PfSPZ of Plasmodium falciparum sporozoite vaccine (PfSPZ-LARC2) vaccine on Days 1, 29, and 57 followed by 3.2x10^3 PfSPZ Challenge (7G8) Controlled Human Malaria Infection (CHMI) on Day 141 administered by direct venous inoculation (DVI). Placebo participants that drop out prior to CHMI will be replaced with infectivity controls. Infectivity controls will receive PfSPZ Challenge (7G8) CHMI N=12
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ (7G8) Challenge
- Group 4 (Placebo Comparator): Healthy malaria-naïve adult participants with no prior history of malaria vaccine study involvement and no exposure to Plasmodium parasites in the past two years, aged between 18 and 45 years will receive saline placebo on Days 1, 29, and 57 followed by 3.2x10^3 PfSPZ Challenge (7G8) Controlled Human Malaria Infection (CHMI) on Day 141 administered by direct venous inoculation (DVI). Placebo participants that drop out prior to CHMI will be replaced with infectivity controls. Infectivity controls will receive PfSPZ Challenge (7G8) CHMI N=6
  Interventions: Biological: PfSPZ (7G8) Challenge; Other: Sodium Chloride, 0.9%

INTERVENTIONS:
Biological: PfSPZ Vaccine — PfSPZ is a candidate vaccine, it consists of a suspension of purified, live-attenuated cryopreserved Pf sporozoites in a cryoprotectant.
  Arms: Group 1; Group 3
Biological: PfSPZ (7G8) Challenge — PfSPZ (7G8) Challenge consists of cryopreserved Plasmodium falciparum (Pf) sporozoites (SPZ) that have been developed to be used to infect volunteers in controlled human malaria infection (CHMI) to assess the efficacy of antimalarial drugs and vaccines. The PfSPZ Challenge (7G8) contains a laboratory malaria clone derived from Brazil.
Other: Sodium Chloride, 0.9% — 0.9% Sodium Chloride Injection
  Arms: Group 2; Group 4

SUMMARY:
This randomized, double-blind, placebo-controlled, Phase 1 trial will enroll up to 22 malaria-naïve, adult participants to test safety, tolerability, immunogenicity, and efficacy of the genetically attenuated Plasmodium falciparum sporozoite vaccine (PfSPZ-LARC2) Vaccine. PfSPZ-LARC2 Vaccine is a late-arresting, replication-competent whole Plasmodium falciparum sporozoite product. We hypothesize that the PfSPZ-LARC2 Vaccine will be safe from breakthrough infection by virtue of deletion of two key parasite genes Mei2 and LINUP and may be more immunogenic and protective than previously tested early arresting sporozoite vaccines. The primary objective is to assess the tolerability and safety of administration of PfSPZ-LARC2 Vaccine, with special attention to the adequacy of attenuation.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, Phase 1 trial will enroll up to 22 malaria-naïve, adult participants to test safety, tolerability, immunogenicity, and efficacy of the genetically attenuated Plasmodium falciparum sporozoite vaccine (PfSPZ-LARC2) Vaccine. PfSPZ-LARC2 Vaccine is a late-arresting, replication-competent whole Plasmodium falciparum sporozoite product. We hypothesize that the PfSPZ-LARC2 Vaccine will be safe from breakthrough infection by virtue of deletion of two key parasite genes Mei2 and LINUP and may be more immunogenic and protective than previously tested early arresting sporozoite vaccines. The vaccine will be produced by Sanaria, Inc. and will be administered by direct venous inoculation (DVI). Placebo control participants will be included in all stages of the study. The study will start with a small set of double-blind, placebo-controlled sentinel participants who will be enrolled first to initially confirm adequate vaccine attenuation before enrolling the remainder of the participants in the study. Vaccine or placebo will be administered three times to participants of the study and then all eligible participants will undergo Controlled Human Malaria Infection (CHMI) to measure protective efficacy compared to placebo. All participants who meet the treatment criteria will be treated with a standard dose of Malarone(R) or Coartem(R).

Participants will be observed for adverse events after each PfSPZ-LARC2 Vaccine or placebo administration as follows. Solicited local and systemic Adverse Events (AEs) related to the vaccine will be recorded beginning of the day of first vaccine administration and continuing through six days after each administration. During the vaccination phase, clinical laboratory evaluations for safety will be performed on venous blood with laboratory toxicities will be monitored from the time of first PfSPZ-LARC2 administration through 14 days after the last PfSPZ-LARC2 administration. Unsolicited AEs related to vaccination will be recorded from the time of first PfSPZ-LARC2 administration through 28 days after the last PfSPZ-LARC2 administration. Serious adverse events (SAEs) will be recorded from the time of first PfSPZ-LARC2 administration through the end of study follow up. Participants will also be monitored for possible breakthrough peripheral parasitemia with Plasmodium 18S rRNA qRT-PCR testing and, if any breakthrough infections are detected, solicited systemic AEs related to such breakthrough infections would be recorded from seven days after each PfSPZ-LARC2 administration until 28 days after each administration. Twelve to 16 weeks after the last vaccine administration, all participants who completed any of the vaccinations will undergo CHMI using P. falciparum strain 7G8 using the Sanaria product PfSPZ Challenge (7G8) at a DVI-administered dose of 3.2x103. Participants will be followed for AEs and evidence of blood-stage infection by Plasmodium 18S rRNA RT-PCR for up to 28 days post-CHMI. Participants showing evidence of infection based on the criteria defined in the protocol will be treated using FDA-approved anti-malarial medication. In addition to safety, tolerability, and efficacy analyses, humoral and cellular immunity of the vaccine will also be evaluated. The primary objective is to assess the tolerability and safety of administration of PfSPZ-LARC2 Vaccine, with special attention to the adequacy of attenuation. The secondary objectives are 1) To assess the efficacy of different PfSPZ-LARC2 Vaccine regimens against CHMI using standard CHMI procedures 2) To assess humoral and cell-mediated immune responses to Pf antigens induced by PfSPZ-LARC2 Vaccine administration.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written informed consent prior to the initiation of any study procedures.
2. Able to understand and agrees to adhere to all planned study procedures and be available for all study visits.
3. Male or non-pregnant female, 18 to 45 years of age (inclusive) at time of enrollment.
4. BMI 18.0-35.0 kg/m^2 at screening.
5. Females of childbearing potential* must agree to use or have practiced true abstinence** or use at least one acceptable primary form of contraception***,****,***** Note: These criteria are applicable to females in a heterosexual relationship and child-bearing potential (i.e., the criteria do not apply to participants in a same sex relationship).

   *Not of childbearing potential - post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy, or Essure(R) placement).

   **True abstinence is 100 percent of time no sexual intercourse (male's penis enters the female's vagina). (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception). If true abstinence changes, then participant agrees to use at least one form of acceptable primary contraception.

   ***Acceptable forms of primary contraception include monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more prior to the participant's enrollment visit (Visit 1), intrauterine devices, birth control pills, barrier methods with spermicide and injectable/implantable/insertable hormonal birth control products.
   * Must use at least one acceptable primary form of contraception for at least 30 days prior to the enrollment visit (Visit 1) and at least one acceptable primary form of contraception for 60 days after the last vaccination or until 28 days post-CHMI, whichever is later.

     * If the participant is treated with Coartem(R) (artemether/lumefantrine - second-line anti-malarial treatment in this study), participants must agree to add an additional barrier method of contraception during treatment.
6. Females of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to enrollment.
7. Males of childbearing potential: use condoms with a female partner of childbearing potential from their enrollment visit (Visit 1), to 60 days after last vaccination or 28 days post-Controlled Human Malaria Infection (CHMI), whichever is later.*,**

   *This does not apply to males in an exclusively same-sex relationship.

   **Biological males who are post-pubertal and considered fertile until permanently sterile by bilateral orchiectomy or vasectomy.
8. Male participants agree to refrain from sperm donation from the time of first vaccination until 60 days after the last vaccination or until 28 days post-CHMI, whichever is later.
9. In good health*

   *As determined by medical history and physical examination to evaluate acute or ongoing chronic medical diagnoses/conditions that have been present for at least 90 days, which would affect the assessment of safety of participants. Chronic medical diagnoses/conditions should be stable for the last 60 days (no hospitalizations, ER, or urgent care for condition or need for supplemental oxygen). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis/condition in the 60 days before enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or done for financial reasons, and in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the participating site PI or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Participants may be on chronic or as needed (prn) medications if, in the opinion of the participating site PI or appropriate sub-investigator, they pose no additional risk to participant safety or assessment of reactogenicity and immunogenicity, and do not indicate a worsening of medical diagnosis/condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided the change was not precipitated by deterioration in the chronic medical condition, and there is no anticipated additional risk to the participant or interference with the evaluation of responses to study vaccination.
10. Oral temperature is less than 100.4 degrees F (38 degrees C).
11. Resting pulse, no greater than 100 beats per minute.
12. Systolic BP is </=140 mm Hg.
13. Clinical screening laboratory evaluations (White Blood Cell Count [WBC], Hemoglobin [Hgb], Platelet Count[PLTs], Absolute Neutrophil Count[ANC], Absolute Lymphocyte Count [ALC], Alanine Aminotransferase [ALT], Aspartate Aminotransferase [AST], creatinine, glucose) are within acceptable normal local reference ranges* *A low creatinine, AST, or ALT value below the normal range are acceptable for trial inclusion as such results are not considered to be clinically significant. If laboratory values are within the normal local reference ranges and Grade 1 (mild) grading criteria are met, these abnormal laboratory values are acceptable for trial inclusion if they are not deemed to be clinically significant by the PI and/or medically trained study clinician listed on Form 1572.
14. Must agree to refrain from donating blood or plasma during the study (outside of this study).
15. Willing to refrain from blood donation for 3 years following CHMI.
16. Agree not to travel to a malaria endemic region until 28 days after CHMI.
17. Willing to take anti-malarial medicines if deemed necessary per protocol or at investigator discretion.
18. Passing score on written Assessment of Understanding (minimum passing score of 80 percent required for participation and one repeat testing is allowed if necessary).

Exclusion Criteria:

1. Unable to provide informed consent including inability to pass the test of understanding.
2. Receipt of a malaria vaccine in a prior clinical trial.
3. History of malaria infection within 2 years prior to study participation.
4. History of a splenectomy or sickle cell disease.
5. History of a non-febrile seizures or complex febrile seizures.
6. Current use of systemic immunosuppressant/immunomodulatory pharmacotherapy.
7. Receipt of a live vaccine within 4 weeks of first vaccination or of 3 or more non-live vaccines within 2 weeks of first vaccination.
8. Receipt of a live vaccine within 4 weeks of CHMI for infectivity controls or of 3 or more non-live vaccines within 2 weeks of CHMI for infectivity controls.
9. Females who are breast-feeding, pregnant or planning to become pregnant during the study period.
10. Known allergy to atovaquone-proguanil (Malarone(R)), artemether-lumefantrine (Coartem(R)), or any component of the investigational products.
11. History of anaphylaxis or other life-threatening reaction to a vaccine.
12. Participation in any study of investigational vaccine/drug <4 weeks before enrollment that in the estimation of the site PI might adversely affect safety or data quality.
13. Evidence of increased cardiovascular disease risk (defined as >10 percent five-year risk by non-laboratory method or prior history of myocardial infarction or myocarditis.
14. Plan to participate in another investigational vaccine/drug research during the study.
15. Plan for major surgery between enrollment until 28 days post-CHMI.
16. Current or anticipated use of any drug with anti-malarial activity that would precede or coincide with malaria challenge or vaccination* *Such medications include but are not limited to doxycycline, tetracycline, erythromycin, clindamycin, azithromycin, trimethoprim/sulfamethoxazole, atovaquone, proguanil, pyrimethamine, quinine, tafenoquine, primaquine, artemisinin derivatives, chloroquine and other 4-amino and 8-aminoquinolines.
17. Current or anticipated use of medications known to cause drug reactions with atovaquone-proguanil or artemether-lumefantrine (e.g., cimetidine, metoclopramide, antacids, and kaolin).
18. Current or anticipated use of medications associated with moderate or high risk for prolonging the QT interval*

    * Such medications include but are not limited to quinine, quinidine, halofantrine, mefloquine, procainamide, disopyramideamiodarone, sotalol, pimozide, ziprasidone, tetracycline, doxycycline, fluoroquinolone, imidazole, and triazole antifungal agents.
19. Current or anticipated use of medications that undergo clinically significant metabolism via the cytochrome enzyme CYP2D6.*

    *Such medications include but are not limited to primaquine, tafenoquine, flecainide, imipramine, amitriptyline, clomipramine.
20. Current or anticipated use of medications that undergo clinically significant metabolism via CYP3A4 or are clinically significant inhibitors or strong inducers of CYP3A4.*,**

    *Such medications include but not limited to (e.g., rifampin, carbamazepine, phenytoin, and/or St. John's wort)

    **Sex hormones, including hormonal contraceptives, are permitted medications.
21. Current or anticipated use of medications that have a clinically significant mixed effect on CYP3A4 (e.g., ritonavir, efavirenz).
22. Known disturbances of the electrolyte balance (e.g., hypokalemia or hypomagnesemia).
23. Positive human immunodeficiency virus (HIV) or hepatitis B surface antigen (HbsAg) serology, or hepatitis C virus (HCV) seropositivity with evidence of HCV viremia.
24. Positive Plasmodium 18S rRNA Reverse Transcription Polymerase Chain Reaction (RT-PCR) at baseline.
25. An abnormal electrocardiogram*

    * An abnormal ECG is defined as one showing pathologic Q waves and significant ST-T wave changes; prolonged QT interval; left ventricular hypertrophy; any non-sinus rhythm including isolated premature ventricular contractions, but excluding isolated premature atrial contractions; right or left bundle branch block; or advanced (secondary or tertiary) A-V heart block; or other clinically significant abnormalities on the electrocardiogram as determined by study clinicians licensed to make medical decisions on the Form FDA 1572.
26. History or family history of prolongation of the QT interval.
27. Any other exclusionary medical, psychiatric, social, behavioral or occupational condition or situation as judged by the site PI intended to ensure participant safety and quality of the trial* *These kind of exclusionary medical, psychiatric, social, behavioral or occupational condition(s) or situation(s) (including active alcohol or drug abuse) include aspects that could impair the participant's ability to give informed consent, increase the risk to the participant of participation in the study, affect the ability of the participant to participate fully in the study, or negatively impact the quality, consistency, integrity or interpretation of data derived from their participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2025-07-23 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Grade 3 laboratory toxicities related to vaccination | Through 14 days after the last vaccination
Occurrence of serious adverse events (SAEs) considered related to vaccination | Through 180 days post-CHMI
Occurrence of solicited local adverse events (AEs) related to the vaccine | Through 6 days after each vaccination
Occurrence of solicited systemic adverse events (AEs) related to the vaccine | Through 6 days after each vaccination
Occurrence of unsolicited adverse events (AEs) considered related to vaccination | Through 28 days after the last vaccination
Proportion of participants with breakthrough blood-stage infection | Through 28 days after last vaccination
  defined as two positive qRT-PCR assays with at least one parasite density of >/=250 estimated parasites/mL from blood samples obtained at least six hours apart or a positive Thick Blood Smear (TBS)
Solicited systemic adverse event (AE) related to the breakthrough infections | Through 28 days after each vaccination

SECONDARY OUTCOMES:
Median Net Optical Density (OD) 1.0 IgG antibodies to Plasmodium falciparum Circumsporozoite Protein (PfCSP) | Up to 16 weeks post-vaccination
  Measured by Enzyme-Linked Immunosorbent Assay (ELISA) on serum samples collected at baseline and post-vaccination prior to Controlled Human Malaria Infection (CHMI)
Percentage of malaria specific CD4+, CD8+, and gamma delta T cells expressing IFN-gamma and/or IL-2 | Up to 16 weeks post-vaccination
  Measured by flow cytometry in PBMCs collected at baseline and post-vaccination prior to Controlled Human Malaria Infection (CHMI)
Proportion of participants with Malaria infection following Controlled Human Malaria Infection (CHMI) | Through 28 days following Controlled Human Malaria Infection (CHMI)
  defined as a two positive qRT-PCR assays of any density taken >/= 6 hours apart, or a positive qRT-PCR assay with a parasite density of >/=250 estimated parasites/mL, or a positive Thick Blood Smear (TBS), on a blood sample

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Washington - Virology Research Clinic, Seattle, Washington, United States

DOCUMENTS (1):
  • Informed Consent Form (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT06735209/ICF_001.pdf